CLINICAL TRIAL: NCT04953559
Title: Transcranial Magnetic Stimulation of the Default Mode Network to Improve Sleep
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Arizona (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 2007900971; W81XWH-19-PRMRP-DA (Other Grant/Funding Number: Department of Defense)
Record Dates: First submitted 2021-04-26; First posted 2021-07-08 (Actual); Last update posted 2022-08-17 (Actual); Status verified 2022-08

CONDITIONS: Insomnia, Primary
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Active cTBS first, then sham cTBS (Experimental): Participants complete an Enrollment Visit followed by one week of at-home actigraphy. Participants return to the lab for Overnight Visit 1 and undergo a MRI scan followed by active cTBS and then another MRI scan followed by a night of polysomnographic monitored in-lab sleep. Participants return home and complete another week of at-home actigraphy. Participants then return to the lab for Overnight Visit 2 where they undergo a MRI scan followed by sham cTBS and then another MRI scan followed by a night of polysomnographic monitored in-lab sleep.
  Interventions: Device: Active cTBS; Device: Sham cTBS
- Sham cTBS first, then active cTBS (Experimental): Participants complete an Enrollment Visit followed by one week of at-home actigraphy. Participants return to the lab for Overnight Visit 1 and undergo a MRI scan followed by sham cTBS and then another MRI scan followed by a night of polysomnographic monitored in-lab sleep. Participants return home and complete another week of at-home actigraphy. Participants then return to the lab for Overnight Visit 2 where they undergo a MRI scan followed by active cTBS and then another MRI scan followed by a night of polysomnographic monitored in-lab sleep.
  Interventions: Device: Active cTBS; Device: Sham cTBS

INTERVENTIONS:
Device: Active cTBS — Active continuous theta burst (cTBS) transcranial magnetic stimulation (TMS)
Device: Sham cTBS — Sham continuous theta burst (cTBS) transcranial magnetic stimulation (TMS)

SUMMARY:
Insomnia is generally believed to be caused by excessive arousal of the brain and body. Rather than transitioning normally and quickly from wakefulness to sleep, individuals with insomnia tend to enter into a self-perpetuating cycle of self-referential thought and arousal. Brain imaging research has shown that these same internally focused self-reflective thoughts tend to activate a core system in the brain known as the Default Mode Network (DMN). The DMN is usually active when a person is internally focused, such as during daydreaming or mind wandering, but tends to be deactivated when the brain is focused on the external environment. The investigators hypothesize that excess activation and connectivity of this brain network may perpetuate internal conversations, worry, and rumination, preventing individuals with insomnia from falling asleep quickly and remaining asleep. Therefore, the goal of the present study is to use a brain stimulation technique known as transcranial magnetic stimulation (TMS) to target the DMN and slightly reduce its activation before bed. This should result in an easier time falling asleep.

For this study, the investigators will recruit 20 healthy individuals and have them sleep in the lab on two occasions. On one occasion, they will be stimulated with a type of TMS called continuous theta burst stimulation (cTBS), which will be targeted toward their DMN. They will then try to sleep in the lab while the investigators record their brain waves using a technique known as polysomnography (PSG). On the other occasion, these same individuals will undergo the same procedure, but the TMS machine will be in a deactivated mode to present a "sham" stimulation. Participants will again try to sleep in the lab following the sham treatment while being recorded with PSG. Neither the participants nor the experimenters will know which condition the participant is receiving at the time. This will only be revealed later. Additionally, all participants will receive a brain scan just before and just after the TMS procedures so that the investigators can examine changes in brain connectivity and chemistry. The investigators expect that the participants will sleep better following the cTBS than following the sham condition and that this will be associated with measurable differences in their brain connectivity and brain chemistry.

If effective, this project would have identified an innovative and novel approach for improving sleep without using drugs.

DETAILED DESCRIPTION:
Individuals with psychophysiological insomnia show greater waking functional connectivity within the DMN compared to healthy individuals. It has been postulated that excessive activation and connectivity of the DMN may be associated with ruminative thinking and internally generated arousal, which makes it difficult to fall asleep.

Primary Objective. The overall objective of this proposal is to temporarily alter the strength of connectivity within the DMN using cTBS before sleep and determine the effects on subsequent sleep. This project is expected to yield robust preliminary data that would allow more extensive research, including a larger follow-on clinical trial to determine the effectiveness of this approach for improving sleep difficulties in military personnel.

The objective of this project will be accomplished through the following Specific Aim:

Specific Aim 1: Determine the effects of cTBS targeted to the DMN on sleep quality, brain neurochemistry, functional connectivity, and next-day cognitive performance.

The investigators' working hypothesis is that relative to sham treatment, cTBS will suppress neural activity within the DMN, leading to improvements in polysomnographically (PSG) measured sleep parameters, and this will be associated with neurochemistry changes and functional connectivity in the DMN, and will improve next day cognitive performance.

Upon completion of this Specific Aim, the expected outcome is to have determined the effects of cTBS on sleep quality, timing, and duration, and identified the brain systems and neurochemistry profiles associated with this change. If successful, this would represent proof-of-concept of a potentially safe non-pharmacologic method to facilitate sleep, and this information could form the basis for follow-on research to refine and further validate this technique to potentially optimize sleep under a variety of militarily-relevant situations.

Insomnia is reported as the most common sleep disorder. It can range in severity, but the most common symptom is difficulty maintaining sleep. Other manifestations of insomnia include early-morning awakenings, and difficulty falling asleep. According to other research, its prevalence is 10 to 15% depending on diagnostic criteria. Roughly 50% of people reporting insomnia have more severe symptoms that meet the criteria for insomnia disorder. Insomnia is conceptualized as a disorder of nocturnal and daytime hyperarousal. This state of arousal is both a cause and a consequence of insomnia. Insomnia causes symptoms that effect people on a cognitive, emotional, and physiological level. People with insomnia often report the feeling of excessive worrying, racing thoughts, and selective attention. Physiologically, insomnia is associated with increased whole-body metabolic rate, increased cortisol levels, increased blood pressure, and elevated brain glucose consumption during both waking and sleeping states. The stressors of chronic insomnia are also associated with an increased risk of developing psychological disorders such as depression and anxiety disorders.

A large number of military personnel report significant sleep difficulties or chronic sleep restriction. In fact, about 42% of military personnel regularly obtain five hours of sleep or less per night, a level that is insufficient to sustain optimal alertness, vigilance, and decision-making. It has been reported that up to 85% of military Service members meet the criteria for a clinically relevant sleep disorder, with approximately 25% having a primary complaint of insomnia (i.e., difficulty falling or staying asleep). Pharmacologic sleep medications may be effective in some situations, but may also be contraindicated in operational environments where alertness is integral. Because sleep problems are among the top complaints of military personnel and can have profound impacts on force readiness, it is imperative that novel approaches to minimizing insomnia and sleep problems be developed.

TMS is a brain stimulation technique which poses far fewer safety risks and adverse experiences than its predecessor, electroconvulsive therapy. TMS has been Food and Drug Administration (FDA)-approved and found effective for use in cases of treatment resistant depression, but has also been utilized off-label to treat OCD and other psychiatric disorders. TMS has demonstrated superior efficacy in the treatment of primary insomnia than both typical medication or psychotherapy treatments. In addition, TMS of the right parietal lobe was shown to be effective for alleviating symptoms of comorbid anxiety and insomnia.

In lay terms, TMS works by targeting electromagnetic fields at particular brain areas from outside of the body. These electromagnetic fields create a current in the brain via the electrochemical firing of brain cells (neurons). This process can influence the function of the targeted brain areas by either facilitating or impairing functional connectivity in a particular network of interconnected brain regions, such as the network associated with daydreaming and self-referential thought (DMN).

The form of TMS to be utilized in present study, continuous theta burst (cTBS), allows for the induction of temporary inhibition of cortical activity using a much shorter length of stimulation as compared to rTMS (repetitive transcranial magnetic stimulation). This protocol was selected for its ability to inhibit, rather than stimulate, activity in the DMN. Prior research using cTBS has shown that this technique can safely and temporarily impair function and connectivity in targeted brain areas. Therefore, the investigators hypothesize that a mild disruption of DMN activation using cTBS prior to sleep will facilitate sleep onset among individuals meeting criteria for primary insomnia, and the investigators further propose that this change will be associated with measurable changes in DMN connectivity and neurochemistry. To test this hypothesis, the investigators will stimulate a node of the DMN approximately two hours before bedtime using cTBS in order to reduce activation and connectivity within the stimulated regions.

ELIGIBILITY:
Inclusion Criteria:

* Healthy men and non-pregnant, non-lactating women 18-50 (inclusive) years of age, free from contraindicated diseases, medications, devices, and conditions.
* Participants must meet the criteria for primary insomnia as determined by scores on the ISI, PSQI, and ESS. Participants must obtain two out of three of the following required scores for each questionnaire:

  * Greater than or equal to 15 for ISI (Gagnon, Belanger, Ivers, & Morin, 2013)
  * Greater than or equal to 6 for PSQI (Buysse et al 1989)
  * Greater than or equal to 11 for ESS (Johns, 2000)

Exclusion Criteria:

* Presence of any metal implant or medical device which may pose a safety risk for MRI or TMS (see below for examples)

  * Cardiac pacemakers
  * Metal clips on blood vessels (also called stents)
  * Artificial heart valves
  * Artificial arms, hands, legs, etc.
  * Brain stimulator devices
  * Implanted drug pumps
  * Ear implants
  * Eye implants or known metal fragments in eyes
  * Exposure to shrapnel or metal filings (wounded in military combat, sheet metal workers, welders, and others)
  * Other metallic surgical hardware in vital areas
  * Certain tattoos with metallic ink
  * Certain transdermal (skin) patches such as NicoDerm (nicotine for tobacco dependence), Transderm Scop (scopolamine for motion sickness), or Ortho Evra (birth control)
* Past or present history of sleep or breathing-related disorders such as sleep apnea (exclusion upon obtaining a score of 3 or higher on the STOP-BANG questionnaire)
* Travel outside the time zone within the two weeks prior to enrollment visit and at any point while active in the study
* Self-reported major medical problems including past or present history of heart problems and/or neurological problems (to include but not limited to heart murmur, heart attack, TBI, stroke, tumor, epilepsy or another seizure disorder)
* Self-reported past or present history of cardiovascular disease (to include but not limited to arrhythmias, valvular heart disease, congestive heart failure, history of sudden cardiac death or myocardial infarction)
* Self-reported past or present history of neurological disorder (to include but not limited to traumatic brain injury including concussions, strokes, tumors, epilepsy or another seizure disorder, amnesia for any reason, hydrocephalus, multiple sclerosis)
* Self-reported past or present history of any seizures or seizure disorders
* Self-reported first-degree family history (like a mother, father, or sibling) of a seizure or seizure disorder
* Self-reported underlying acute or chronic pulmonary disease requiring daily inhaler use
* Self-reported history of fainting spells or syncope
* Self-reported past (at any point in the participant's history) or present psychiatric problems not including depression and/or anxiety disorders (to include but not limited to bipolar, mania, ADHD, or psychotic disorders)
* Self-reported history of depression and/or anxiety disorders within the past 2 years
* Self-reported suicidal ideation as indicated by a score equal to or greater than 2 on the BDI
* Self-reported current use of certain prescription medications including Ambien, benzodiazepines, stimulants (amphetamines, medication for narcolepsy), antidepressants (SSRIs, SNRIs), antipsychotics, blood pressure medications, thyroid medications.
* Self-reported current use of supplements that may affect sleep (to include but not limited to melatonin, valerian root, kava root)
* Self-reported caffeine use in excess of 300 mg (e.g., approximately 8 caffeinated sodas or approximately 3-4 12-oz cups of coffee) per day on average
* Self-reported or suspected regular nicotine use (or addiction) (defined as more than 1 cigarette or equivalent per week within the last 1 year)
* Self-reported or suspected heavy alcohol use (minimum limit to define heavy alcohol use is 14 drinks per week)
* Self-reported or suspected use of illicit drugs (to include but not limited to benzodiazepines, amphetamines, cocaine, opioids)
* (Females only) Positive urine pregnancy result (Urine HCG Test results)
* (Females only) Self-reported or suspected current breast-feeding or collecting breast-milk
* Learned English past age 3
* Speaking English as a non-primary language
* Less than 9th grade education
* Unusual sleep schedules in past six months
* Overnight shift work
* Inability to read and sign consent
* Failure to cooperate with requirements of the study

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2021-08-06 (Actual); Primary Completion 2022-08-31 (Estimated); Study Completion 2022-08-31 (Estimated)

PRIMARY OUTCOMES:
Within-subject changes in functional connectivity and brain metabolites following administration of active or sham cTBS TMS - day 8 | Once during Overnight Visit 1 pre-TMS MRI scan session (day 8)
  Measure neurochemistry in anterior cingulate and occipitoparietal cortex using spectroscopy during MRI scan
Within-subject changes in functional connectivity and brain metabolites following administration of active or sham cTBS TMS - day 8 | Once during Overnight Visit 1 post-TMS MRI scan session (day 8)
  Measure neurochemistry in anterior cingulate and occipitoparietal cortex using spectroscopy during MRI scan
Within-subject changes in functional connectivity and brain metabolites following administration of active or sham cTBS TMS - day 15 | Once during Overnight Visit 2 pre-TMS MRI scan session (day 15)
  Measure neurochemistry in anterior cingulate and occipitoparietal cortex using spectroscopy during MRI scan
Within-subject changes in functional connectivity and brain metabolites following administration of active or sham cTBS TMS - day 15 | Once during Overnight 2 post-TMS MRI scan session (day 15)
  Measure neurochemistry in anterior cingulate and occipitoparietal cortex using spectroscopy during MRI scan
Sleep onset latency (SOL) following administration of active or sham cTBS TMS - day 8 | During in-lab periods while sleeping during Overnight Visit 1 (day 8-9)
  Sleep period polysomnographic (PSG) measurement
Sleep onset latency (SOL) following administration of active or sham cTBS TMS | During in-lab periods while sleeping during Overnight Visit 2 (day 15-16)
  Sleep period polysomnographic (PSG) measurement day 15
Total sleep time (TST) following administration of active or sham cTBS TMS - day 8-9 | During in-lab periods while sleeping during Overnight Visit 1 (day 8-9)
  Sleep period polysomnographic (PSG) measurement
Total sleep time (TST) following administration of active or sham cTBS TMS - day 15-16 | During in-lab periods while sleeping during Overnight Visit 2 (day 15-16)
  Sleep period polysomnographic (PSG) measurement
Sleep efficiency (SE) following administration of active or sham cTBS TMS - day 8-9 | During in-lab periods while sleeping during Overnight Visit 1 (day 8-9)
  Sleep period polysomnographic (PSG) measurement
Sleep efficiency (SE) following administration of active or sham cTBS TMS - day 8-9 | During in-lab periods while sleeping during Overnight Visit 2 (day 15-16)
  Sleep period polysomnographic (PSG) measurement
Wake after sleep onset (WASO) following administration of active or sham cTBS TMS - day 8-9 | During in-lab periods while sleeping during Overnight Visit 1 (day 8-9)
  Sleep period polysomnographic (PSG) measurement
Wake after sleep onset (WASO) following administration of active or sham cTBS TMS - day 15-16 | During in-lab periods while sleeping during Overnight Visit 2 (day 15-16)
  Sleep period polysomnographic (PSG) measurement
Time spent in each sleep stage following administration of active or sham cTBS TMS | During in-lab periods while sleeping during Overnight Visit 1 (day 8-9)
  Sleep period polysomnographic (PSG) measurement (time) day 8
Percentage of time spent in each sleep stage following administration of active or sham cTBS TMS | During in-lab periods while sleeping during Overnight Visit 1 (day 8-9)
  Sleep period polysomnographic (PSG) measurement (percentage of time) day 8
Time spent in each sleep stage following administration of active or sham cTBS TMS | During in-lab periods while sleeping during Overnight Visit 2 (day 15-16)
  Sleep period polysomnographic (PSG) measurement (time) day 15
Percentage of time spent in each sleep stage following administration of active or sham cTBS TMS | During in-lab periods while sleeping during Overnight Visit 2 (day 15-16)
  Sleep period polysomnographic (PSG) measurement (percentage of time) day 15

SECONDARY OUTCOMES:
Karolinska Sleepiness Scale (KSS) - day 8, admin 1 | Once during cognitive testing portion of Overnight Visit 1 (day 8-9), day 8
  To evaluate effects of sleep schedule on subjective sleepiness. Volunteers are presented with a 9-point sleepiness scale on a computer monitor (1=very alert, 3=alert, 5=neither alert nor sleepy, 7=sleepy (but not fighting sleep), 9=very sleepy (fighting sleep) and select the number on the scale that best reflects their current level of subjective sleepiness.
Karolinska Sleepiness Scale (KSS) - day 8, admin 2 | Approximately one hour after previous administration during cognitive testing portion of Overnight Visit 1 (day 8-9), day 8
  To evaluate effects of sleep schedule on subjective sleepiness. Volunteers are presented with a 9-point sleepiness scale on a computer monitor (1=very alert, 3=alert, 5=neither alert nor sleepy, 7=sleepy (but not fighting sleep), 9=very sleepy (fighting sleep) and select the number on the scale that best reflects their current level of subjective sleepiness.
Karolinska Sleepiness Scale (KSS) - day 8, admin 3 | Approximately one hour after previous administration (2 hours after initial) during cognitive testing portion of Overnight Visit 1 (day 8-9), day 8
  To evaluate effects of sleep schedule on subjective sleepiness. Volunteers are presented with a 9-point sleepiness scale on a computer monitor (1=very alert, 3=alert, 5=neither alert nor sleepy, 7=sleepy (but not fighting sleep), 9=very sleepy (fighting sleep) and select the number on the scale that best reflects their current level of subjective sleepiness.
Karolinska Sleepiness Scale (KSS) - day 9, admin 4 | Once during cognitive testing portion of Overnight Visit 1 (day 8-9), day 9
  To evaluate effects of sleep schedule on subjective sleepiness. Volunteers are presented with a 9-point sleepiness scale on a computer monitor (1=very alert, 3=alert, 5=neither alert nor sleepy, 7=sleepy (but not fighting sleep), 9=very sleepy (fighting sleep) and select the number on the scale that best reflects their current level of subjective sleepiness.
Karolinska Sleepiness Scale (KSS) - day 9, admin 5 | Approximately one hour after previous administration during cognitive testing portion of Overnight Visit 1 (day 8-9), day 9
  To evaluate effects of sleep schedule on subjective sleepiness. Volunteers are presented with a 9-point sleepiness scale on a computer monitor (1=very alert, 3=alert, 5=neither alert nor sleepy, 7=sleepy (but not fighting sleep), 9=very sleepy (fighting sleep) and select the number on the scale that best reflects their current level of subjective sleepiness.
Karolinska Sleepiness Scale (KSS) - day 9, admin 6 | Approximately one hour after previous administration (2 hours after initial) during cognitive testing portion of Overnight Visit 1 (day 8-9), day 9
  To evaluate effects of sleep schedule on subjective sleepiness. Volunteers are presented with a 9-point sleepiness scale on a computer monitor (1=very alert, 3=alert, 5=neither alert nor sleepy, 7=sleepy (but not fighting sleep), 9=very sleepy (fighting sleep) and select the number on the scale that best reflects their current level of subjective sleepiness.
Karolinska Sleepiness Scale (KSS) - day 15, admin 1 | Once during cognitive testing portion of Overnight Visit 2 (day 15-16), day 15
  To evaluate effects of sleep schedule on subjective sleepiness. Volunteers are presented with a 9-point sleepiness scale on a computer monitor (1=very alert, 3=alert, 5=neither alert nor sleepy, 7=sleepy (but not fighting sleep), 9=very sleepy (fighting sleep) and select the number on the scale that best reflects their current level of subjective sleepiness.
Karolinska Sleepiness Scale (KSS) - day 15, admin 2 | Approximately one hour after previous administration during cognitive testing portion of Overnight Visit 2 (day 15-16), day 15
  To evaluate effects of sleep schedule on subjective sleepiness. Volunteers are presented with a 9-point sleepiness scale on a computer monitor (1=very alert, 3=alert, 5=neither alert nor sleepy, 7=sleepy (but not fighting sleep), 9=very sleepy (fighting sleep) and select the number on the scale that best reflects their current level of subjective sleepiness.
Karolinska Sleepiness Scale (KSS) - day 15, admin 3 | Approximately one hour after previous administration (2 hours after initial) during cognitive testing portion of Overnight Visit 2 (day 15-16), day 15
  To evaluate effects of sleep schedule on subjective sleepiness. Volunteers are presented with a 9-point sleepiness scale on a computer monitor (1=very alert, 3=alert, 5=neither alert nor sleepy, 7=sleepy (but not fighting sleep), 9=very sleepy (fighting sleep) and select the number on the scale that best reflects their current level of subjective sleepiness.
Karolinska Sleepiness Scale (KSS) - day 16, admin 4 | Once during cognitive testing portion of Overnight Visit 2 (day 15-16), day 16
  To evaluate effects of sleep schedule on subjective sleepiness. Volunteers are presented with a 9-point sleepiness scale on a computer monitor (1=very alert, 3=alert, 5=neither alert nor sleepy, 7=sleepy (but not fighting sleep), 9=very sleepy (fighting sleep) and select the number on the scale that best reflects their current level of subjective sleepiness.
Karolinska Sleepiness Scale (KSS) - day 16, admin 5 | Approximately one hour after previous administration during cognitive testing portion of Overnight Visit 2 (day 15-16), day 16
  To evaluate effects of sleep schedule on subjective sleepiness. Volunteers are presented with a 9-point sleepiness scale on a computer monitor (1=very alert, 3=alert, 5=neither alert nor sleepy, 7=sleepy (but not fighting sleep), 9=very sleepy (fighting sleep) and select the number on the scale that best reflects their current level of subjective sleepiness.
Karolinska Sleepiness Scale (KSS) - day 16, admin 6 | Approximately one hour after previous administration (2 hours after initial) during cognitive testing portion of Overnight Visit 2 (day 15-16), day 16
  To evaluate effects of sleep schedule on subjective sleepiness. Volunteers are presented with a 9-point sleepiness scale on a computer monitor (1=very alert, 3=alert, 5=neither alert nor sleepy, 7=sleepy (but not fighting sleep), 9=very sleepy (fighting sleep) and select the number on the scale that best reflects their current level of subjective sleepiness.
Psychomotor Vigilance Tests (PVT) - day 1, admin 1 (mean RT) | Once during cognitive testing on Enrollment day (day 1)
  To assess the effects of sleep loss on visual reaction time as a behavioral measure of sleepiness, participants continuously monitor a blank display and click a keyboard button as quickly as possible in response to a visual stimulus (i.e. an "X" that appears on the computer screen). Mean RT (ms)
Psychomotor Vigilance Tests (PVT) - day 1, admin 1 (mean Speed) | Once during cognitive testing on Enrollment day (day 1)
  To assess the effects of sleep loss on visual reaction time as a behavioral measure of sleepiness, participants continuously monitor a blank display and click a keyboard button as quickly as possible in response to a visual stimulus (i.e. an "X" that appears on the computer screen). Mean Speed (s-1)
Psychomotor Vigilance Tests (PVT) - day 1, admin 1 (Lapses) | Once during cognitive testing on Enrollment day (day 1)
  To assess the effects of sleep loss on visual reaction time as a behavioral measure of sleepiness, participants continuously monitor a blank display and click a keyboard button as quickly as possible in response to a visual stimulus (i.e. an "X" that appears on the computer screen). Lapses (#)
Psychomotor Vigilance Tests (PVT) - day 1, admin 2 (mean RT) | Approximately one hour after previous administration during cognitive testing on Enrollment day (day 1)
  To assess the effects of sleep loss on visual reaction time as a behavioral measure of sleepiness, participants continuously monitor a blank display and click a keyboard button as quickly as possible in response to a visual stimulus (i.e. an "X" that appears on the computer screen). Mean RT (ms)
Psychomotor Vigilance Tests (PVT) - day 1, admin 2 (mean Speed) | Approximately one hour after previous administration during cognitive testing on Enrollment day (day 1)
  To assess the effects of sleep loss on visual reaction time as a behavioral measure of sleepiness, participants continuously monitor a blank display and click a keyboard button as quickly as possible in response to a visual stimulus (i.e. an "X" that appears on the computer screen). Mean Speed (s-1)
Psychomotor Vigilance Tests (PVT) - day 1, admin 2 (Lapses) | Approximately one hour after previous administration during cognitive testing on Enrollment day (day 1)
  To assess the effects of sleep loss on visual reaction time as a behavioral measure of sleepiness, participants continuously monitor a blank display and click a keyboard button as quickly as possible in response to a visual stimulus (i.e. an "X" that appears on the computer screen). Lapses (#)
Psychomotor Vigilance Tests (PVT) - day 8, admin 3 (mean RT) | Once during cognitive testing of Overnight Visit 1 (day 8-9), day 8
  To assess the effects of sleep loss on visual reaction time as a behavioral measure of sleepiness, participants continuously monitor a blank display and click a keyboard button as quickly as possible in response to a visual stimulus (i.e. an "X" that appears on the computer screen). Mean RT (ms)
Psychomotor Vigilance Tests (PVT) - day 8, admin 3 (mean Speed) | Once during cognitive testing of Overnight Visit 1 (day 8-9), day 8
  To assess the effects of sleep loss on visual reaction time as a behavioral measure of sleepiness, participants continuously monitor a blank display and click a keyboard button as quickly as possible in response to a visual stimulus (i.e. an "X" that appears on the computer screen). Mean Speed (s-1)
Psychomotor Vigilance Tests (PVT) - day 8, admin 3 (Lapses) | Once during cognitive testing of Overnight Visit 1 (day 8-9), day 8
  To assess the effects of sleep loss on visual reaction time as a behavioral measure of sleepiness, participants continuously monitor a blank display and click a keyboard button as quickly as possible in response to a visual stimulus (i.e. an "X" that appears on the computer screen). Lapses (#)
Psychomotor Vigilance Tests (PVT) - day 15, admin 9 (mean RT) | Once during cognitive testing of Overnight Visit 2 (day 15)
  To assess the effects of sleep loss on visual reaction time as a behavioral measure of sleepiness, participants continuously monitor a blank display and click a keyboard button as quickly as possible in response to a visual stimulus (i.e. an "X" that appears on the computer screen). Mean RT (ms)
Psychomotor Vigilance Tests (PVT) - day 15, admin 9 (mean Speed) | Once during cognitive testing of Overnight Visit 2 (day 15)
  To assess the effects of sleep loss on visual reaction time as a behavioral measure of sleepiness, participants continuously monitor a blank display and click a keyboard button as quickly as possible in response to a visual stimulus (i.e. an "X" that appears on the computer screen). Mean Speed (s-1)
Psychomotor Vigilance Tests (PVT) - day 15, admin 9 (Lapses) | Once during cognitive testing of Overnight Visit 2 (day 15)
  To assess the effects of sleep loss on visual reaction time as a behavioral measure of sleepiness, participants continuously monitor a blank display and click a keyboard button as quickly as possible in response to a visual stimulus (i.e. an "X" that appears on the computer screen). Mean Speed (s-1)
Psychomotor Vigilance Tests (PVT) - day 8, admin 4 (mean RT) | Approximately one hour after previous administration during cognitive testing of Overnight Visit 1 (day 8-9), day 8
  To assess the effects of sleep loss on visual reaction time as a behavioral measure of sleepiness, participants continuously monitor a blank display and click a keyboard button as quickly as possible in response to a visual stimulus (i.e. an "X" that appears on the computer screen). Mean RT (ms)
Psychomotor Vigilance Tests (PVT) - day 8, admin 4 (mean Speed) | Approximately one hour after previous administration during cognitive testing of Overnight Visit 1 (day 8-9), day 8
  To assess the effects of sleep loss on visual reaction time as a behavioral measure of sleepiness, participants continuously monitor a blank display and click a keyboard button as quickly as possible in response to a visual stimulus (i.e. an "X" that appears on the computer screen). Mean Speed (s-1)
Psychomotor Vigilance Tests (PVT) - day 8, admin 4 (Lapses) | Approximately one hour after previous administration during cognitive testing of Overnight Visit 1 (day 8-9), day 8
  To assess the effects of sleep loss on visual reaction time as a behavioral measure of sleepiness, participants continuously monitor a blank display and click a keyboard button as quickly as possible in response to a visual stimulus (i.e. an "X" that appears on the computer screen). Lapses (#)
Psychomotor Vigilance Tests (PVT) - day 15, admin 10 (mean RT) | Approximately one hour after previous administration during cognitive testing of Overnight Visit 2 (day 15-16), day 15
  To assess the effects of sleep loss on visual reaction time as a behavioral measure of sleepiness, participants continuously monitor a blank display and click a keyboard button as quickly as possible in response to a visual stimulus (i.e. an "X" that appears on the computer screen). Mean RT (ms)
Psychomotor Vigilance Tests (PVT) - day 15, admin 10 (mean Speed) | Approximately one hour after previous administration during cognitive testing of Overnight Visit 2 (day 15-16), day 15
  To assess the effects of sleep loss on visual reaction time as a behavioral measure of sleepiness, participants continuously monitor a blank display and click a keyboard button as quickly as possible in response to a visual stimulus (i.e. an "X" that appears on the computer screen). Mean Speed (s-1)
Psychomotor Vigilance Tests (PVT) - day 15, admin 10 (Lapses) | Approximately one hour after previous administration during cognitive testing of Overnight Visit 2 (day 15-16), day 15
  To assess the effects of sleep loss on visual reaction time as a behavioral measure of sleepiness, participants continuously monitor a blank display and click a keyboard button as quickly as possible in response to a visual stimulus (i.e. an "X" that appears on the computer screen). Lapses (#)
Psychomotor Vigilance Tests (PVT) - day 8, admin 5 (mean RT) | Approximately one hour after previous administration (2 hours after initial) during cognitive testing of Overnight Visit 1 (day 8-9), day 8
  To assess the effects of sleep loss on visual reaction time as a behavioral measure of sleepiness, participants continuously monitor a blank display and click a keyboard button as quickly as possible in response to a visual stimulus (i.e. an "X" that appears on the computer screen). Mean RT (ms)
Psychomotor Vigilance Tests (PVT) - day 8, admin 5 (mean Speed) | Approximately one hour after previous administration (2 hours after initial) during cognitive testing of Overnight Visit 1 (day 8-9), day 8
  To assess the effects of sleep loss on visual reaction time as a behavioral measure of sleepiness, participants continuously monitor a blank display and click a keyboard button as quickly as possible in response to a visual stimulus (i.e. an "X" that appears on the computer screen). Mean Speed (s-1)
Psychomotor Vigilance Tests (PVT) - day 8, admin 5 (Lapses) | Approximately one hour after previous administration (2 hours after initial) during cognitive testing of Overnight Visit 1 (day 8-9), day 8
  To assess the effects of sleep loss on visual reaction time as a behavioral measure of sleepiness, participants continuously monitor a blank display and click a keyboard button as quickly as possible in response to a visual stimulus (i.e. an "X" that appears on the computer screen). Lapses (#)
Psychomotor Vigilance Tests (PVT) - day 15, admin 11 (mean RT) | Approximately one hour after previous administration (2 hours after initial) during cognitive testing of Overnight Visit 2 (day 15-16), day 15
  To assess the effects of sleep loss on visual reaction time as a behavioral measure of sleepiness, participants continuously monitor a blank display and click a keyboard button as quickly as possible in response to a visual stimulus (i.e. an "X" that appears on the computer screen). Mean RT (ms)
Psychomotor Vigilance Tests (PVT) - day 15, admin 11 (mean Speed) | Approximately one hour after previous administration (2 hours after initial) during cognitive testing of Overnight Visit 2 (day 15-16), day 15
  To assess the effects of sleep loss on visual reaction time as a behavioral measure of sleepiness, participants continuously monitor a blank display and click a keyboard button as quickly as possible in response to a visual stimulus (i.e. an "X" that appears on the computer screen). Mean Speed (s-1)
Psychomotor Vigilance Tests (PVT) - day 15, admin 11 (Lapses) | Approximately one hour after previous administration (2 hours after initial) during cognitive testing of Overnight Visit 2 (day 15-16), day 15
  To assess the effects of sleep loss on visual reaction time as a behavioral measure of sleepiness, participants continuously monitor a blank display and click a keyboard button as quickly as possible in response to a visual stimulus (i.e. an "X" that appears on the computer screen). Lapses (#)
Psychomotor Vigilance Tests (PVT) - day 9, admin 6 (mean RT) | Once during cognitive testing during Overnight Visit 1 (day 8-9), day 9
  To assess the effects of sleep loss on visual reaction time as a behavioral measure of sleepiness, participants continuously monitor a blank display and click a keyboard button as quickly as possible in response to a visual stimulus (i.e. an "X" that appears on the computer screen). Mean RT (ms)
Psychomotor Vigilance Tests (PVT) - day 9, admin 6 (mean Speed) | Once during cognitive testing during Overnight Visit 1 (day 8-9), day 9
  To assess the effects of sleep loss on visual reaction time as a behavioral measure of sleepiness, participants continuously monitor a blank display and click a keyboard button as quickly as possible in response to a visual stimulus (i.e. an "X" that appears on the computer screen). Mean Speed (s-1)
Psychomotor Vigilance Tests (PVT) - day 9, admin 6 (Lapses) | Once during cognitive testing during Overnight Visit 1 (day 8-9), day 9
  To assess the effects of sleep loss on visual reaction time as a behavioral measure of sleepiness, participants continuously monitor a blank display and click a keyboard button as quickly as possible in response to a visual stimulus (i.e. an "X" that appears on the computer screen). Lapses (#)
Psychomotor Vigilance Tests (PVT) - day 16, admin 12 (mean RT) | Once during cognitive testing during Overnight Visit 2 (day 15-16), day 16
  To assess the effects of sleep loss on visual reaction time as a behavioral measure of sleepiness, participants continuously monitor a blank display and click a keyboard button as quickly as possible in response to a visual stimulus (i.e. an "X" that appears on the computer screen). Mean RT (ms)
Psychomotor Vigilance Tests (PVT) - day 16, admin 12 (mean Speed) | Once during cognitive testing during Overnight Visit 2 (day 15-16), day 16
  To assess the effects of sleep loss on visual reaction time as a behavioral measure of sleepiness, participants continuously monitor a blank display and click a keyboard button as quickly as possible in response to a visual stimulus (i.e. an "X" that appears on the computer screen). Mean Speed (s-1)
Psychomotor Vigilance Tests (PVT) - day 16, admin 12 (Lapses) | Once during cognitive testing during Overnight Visit 2 (day 15-16), day 16
  To assess the effects of sleep loss on visual reaction time as a behavioral measure of sleepiness, participants continuously monitor a blank display and click a keyboard button as quickly as possible in response to a visual stimulus (i.e. an "X" that appears on the computer screen). Lapses (#)
Psychomotor Vigilance Tests (PVT) - day 9, admin 7 (mean Speed) | Approximately one hour after previous administration during cognitive testing of Overnight Visit 1 (day 8-9), day 9
  To assess the effects of sleep loss on visual reaction time as a behavioral measure of sleepiness, participants continuously monitor a blank display and click a keyboard button as quickly as possible in response to a visual stimulus (i.e. an "X" that appears on the computer screen). Mean Speed (s-1)
Psychomotor Vigilance Tests (PVT) - day 9, admin 7 (mean RT) | Approximately one hour after previous administration during cognitive testing of Overnight Visit 1 (day 8-9), day 9
  To assess the effects of sleep loss on visual reaction time as a behavioral measure of sleepiness, participants continuously monitor a blank display and click a keyboard button as quickly as possible in response to a visual stimulus (i.e. an "X" that appears on the computer screen). Mean RT (ms)
Psychomotor Vigilance Tests (PVT) - day 9, admin 7 (Lapses) | Approximately one hour after previous administration during cognitive testing of Overnight Visit 1 (day 8-9), day 9
  To assess the effects of sleep loss on visual reaction time as a behavioral measure of sleepiness, participants continuously monitor a blank display and click a keyboard button as quickly as possible in response to a visual stimulus (i.e. an "X" that appears on the computer screen). Lapses (#)
Psychomotor Vigilance Tests (PVT) - day 16, admin 12 (mean RT) | Approximately one hour after previous administration during cognitive testing of Overnight Visit 2 (day 15-16), day 16
  To assess the effects of sleep loss on visual reaction time as a behavioral measure of sleepiness, participants continuously monitor a blank display and click a keyboard button as quickly as possible in response to a visual stimulus (i.e. an "X" that appears on the computer screen). Mean RT (ms)
Psychomotor Vigilance Tests (PVT) - day 16, admin 12 (mean Speed) | Approximately one hour after previous administration during cognitive testing of Overnight Visit 2 (day 15-16), day 16
  To assess the effects of sleep loss on visual reaction time as a behavioral measure of sleepiness, participants continuously monitor a blank display and click a keyboard button as quickly as possible in response to a visual stimulus (i.e. an "X" that appears on the computer screen). Mean Speed (s-1)
Psychomotor Vigilance Tests (PVT) - day 16, admin 12 (Lapses) | Approximately one hour after previous administration during cognitive testing of Overnight Visit 2 (day 15-16), day 16
  To assess the effects of sleep loss on visual reaction time as a behavioral measure of sleepiness, participants continuously monitor a blank display and click a keyboard button as quickly as possible in response to a visual stimulus (i.e. an "X" that appears on the computer screen). Lapses (#)
Psychomotor Vigilance Tests (PVT) - day 9, admin 8 (mean RT) | Approximately one hour after previous administration (2 hours after initial) during cognitive testing of Overnight Visit 1 (day 8-9), day 9
  To assess the effects of sleep loss on visual reaction time as a behavioral measure of sleepiness, participants continuously monitor a blank display and click a keyboard button as quickly as possible in response to a visual stimulus (i.e. an "X" that appears on the computer screen). Mean RT (ms)
Psychomotor Vigilance Tests (PVT) - day 9, admin 8 (mean Speed) | Approximately one hour after previous administration (2 hours after initial) during cognitive testing of Overnight Visit 1 (day 8-9), day 9
  To assess the effects of sleep loss on visual reaction time as a behavioral measure of sleepiness, participants continuously monitor a blank display and click a keyboard button as quickly as possible in response to a visual stimulus (i.e. an "X" that appears on the computer screen). Mean Speed (s-1)
Psychomotor Vigilance Tests (PVT) - day 9, admin 8 (Lapses) | Approximately one hour after previous administration (2 hours after initial) during cognitive testing of Overnight Visit 1 (day 8-9), day 9
  To assess the effects of sleep loss on visual reaction time as a behavioral measure of sleepiness, participants continuously monitor a blank display and click a keyboard button as quickly as possible in response to a visual stimulus (i.e. an "X" that appears on the computer screen). Lapses (#)
Psychomotor Vigilance Tests (PVT) - day 16, admin 13 (mean RT) | Approximately one hour after previous administration (2 hours after initial) during cognitive testing of Overnight Visit 2 (day 15-16), day 16
  To assess the effects of sleep loss on visual reaction time as a behavioral measure of sleepiness, participants continuously monitor a blank display and click a keyboard button as quickly as possible in response to a visual stimulus (i.e. an "X" that appears on the computer screen). Mean RT (ms)
Psychomotor Vigilance Tests (PVT) - day 16, admin 13 (mean Speed) | Approximately one hour after previous administration (2 hours after initial) during cognitive testing of Overnight Visit 2 (day 15-16), day 16
  To assess the effects of sleep loss on visual reaction time as a behavioral measure of sleepiness, participants continuously monitor a blank display and click a keyboard button as quickly as possible in response to a visual stimulus (i.e. an "X" that appears on the computer screen). Mean Speed (s-1)
Psychomotor Vigilance Tests (PVT) - day 16, admin 13 (Lapses) | Approximately one hour after previous administration (2 hours after initial) during cognitive testing of Overnight Visit 2 (day 15-16), day 16
  To assess the effects of sleep loss on visual reaction time as a behavioral measure of sleepiness, participants continuously monitor a blank display and click a keyboard button as quickly as possible in response to a visual stimulus (i.e. an "X" that appears on the computer screen). Lapses (#)
Spielberger State-Trait Anxiety Inventory - State (STAI-S) - day 1 | During cognitive testing portion of Enrollment Day (day 1)
  Used to identify state changes in anxiety in healthy adults. Volunteers are instructed to rate on a four-point scale how closely they identify with 20 statements related to state anxiety. State anxiety level (20-80), higher scores indicate greater state anxiety.
Spielberger State-Trait Anxiety Inventory - State (STAI-S) - day 8 | During cognitive testing portion of Overnight Visit 1 (day 8)
  Used to identify state changes in anxiety in healthy adults. Volunteers are instructed to rate on a four-point scale how closely they identify with 20 statements related to state anxiety. State anxiety level (20-80), higher scores indicate greater state anxiety.
Spielberger State-Trait Anxiety Inventory - State (STAI-S) - day 15 | During cognitive testing portion of Overnight Visit 2 (day 15)
  Used to identify state changes in anxiety in healthy adults. Volunteers are instructed to rate on a four-point scale how closely they identify with 20 statements related to state anxiety. State anxiety level (20-80), higher scores indicate greater state anxiety.
Actigraphy | Throughout the entire study, except during MRI and TMS administration - up to 14 days
  To determine amount and timing of sleep/wake periods during all phases of the study. Except for epochs that may be removed manually if they are determined to contain artifact, actigraphy records will be automatically scored by computer as either "sleep" or "wake" using the algorithms provided by the various manufacturers. Wear the one actigraph (approximately the size of a diver's wristwatch) continuously across all study phases, including at home.
Glasgow Content of Thoughts Inventory (GCTI) - day 1 | During cognitive testing portion of Enrollment Day (day 1)
  Evaluate the content, character, and intrusiveness of cognitions in the moments prior to sleep onset, specifically in those with insomnia. Rate 25 statements on a scale from 1 ("never") to 4 ("always"). Level of intrusive thoughts prior to sleep (25-100) with higher scores indicating more intrusive cognitions.
Glasgow Content of Thoughts Inventory (GCTI) - day 8 | During cognitive testing portion of Overnight Visit 1 (day 8)
  Evaluate the content, character, and intrusiveness of cognitions in the moments prior to sleep onset, specifically in those with insomnia. Rate 25 statements on a scale from 1 ("never") to 4 ("always"). Level of intrusive thoughts prior to sleep (25-100) with higher scores indicating more intrusive cognitions.
Glasgow Content of Thoughts Inventory (GCTI) - day 15 | During cognitive testing portion of Overnight Visit 2 (day 15)
  Evaluate the content, character, and intrusiveness of cognitions in the moments prior to sleep onset, specifically in those with insomnia. Rate 25 statements on a scale from 1 ("never") to 4 ("always"). Level of intrusive thoughts prior to sleep (25-100) with higher scores indicating more intrusive cognitions.
Visual Analog Mood Scale (VAMS) - day 8, admin 1 | During evening of Overnight Visit 1 (day 8)
  Brief measure of subjective mood. Participants will be presented with eight specific mood states: Afraid, Confused, Sad, Angry, Energetic, Tired, Happy, and Tense. For each scale, a neutral schematic face is at the top of 100mm vertical line, with a mood face at the bottom of the line. Participants draw a line on the scale that best describes how they are currently feeling. Subjective mood for each of eight mood states (Afraid, Confused, Sad, Angry, Energetic, Tired, Happy, and Tense).
Visual Analog Mood Scale (VAMS) - day 9, admin 2 | During morning of Overnight Visit 1 (day 9)
  Brief measure of subjective mood. Participants will be presented with eight specific mood states: Afraid, Confused, Sad, Angry, Energetic, Tired, Happy, and Tense. For each scale, a neutral schematic face is at the top of 100mm vertical line, with a mood face at the bottom of the line. Participants draw a line on the scale that best describes how they are currently feeling. Subjective mood for each of eight mood states (Afraid, Confused, Sad, Angry, Energetic, Tired, Happy, and Tense).
Visual Analog Mood Scale (VAMS) - day 15, admin 1 | During evening of Overnight Visit 2 (day 15)
  Brief measure of subjective mood. Participants will be presented with eight specific mood states: Afraid, Confused, Sad, Angry, Energetic, Tired, Happy, and Tense. For each scale, a neutral schematic face is at the top of 100mm vertical line, with a mood face at the bottom of the line. Participants draw a line on the scale that best describes how they are currently feeling. Subjective mood for each of eight mood states (Afraid, Confused, Sad, Angry, Energetic, Tired, Happy, and Tense).
Visual Analog Mood Scale (VAMS) - day 16, admin 2 | During morning of Overnight Visit 2 (day 16)
  Brief measure of subjective mood. Participants will be presented with eight specific mood states: Afraid, Confused, Sad, Angry, Energetic, Tired, Happy, and Tense. For each scale, a neutral schematic face is at the top of 100mm vertical line, with a mood face at the bottom of the line. Participants draw a line on the scale that best describes how they are currently feeling. Subjective mood for each of eight mood states (Afraid, Confused, Sad, Angry, Energetic, Tired, Happy, and Tense).
California Verbal Learning Test Third Edition (CVLT-3) - day 8-9 | Learn the list and recall the list once during Overnight Visit 1 (day 8-9)
  To assess verbal memory and learning. Volunteers will listen to a series of words during cognitive testing on the first day of their overnight visits. On the second day of their overnight visit, they will be asked to recall the list of words and which category each word belongs to.
California Verbal Learning Test Third Edition (CVLT-3) - day 15-16 | Learn the list and recall the list once during Overnight Visit 2 (day 15-16)
  To assess verbal memory and learning. Volunteers will listen to a series of words during cognitive testing on the first day of their overnight visits. On the second day of their overnight visit, they will be asked to recall the list of words and which category each word belongs to.
Repeatable Battery for Neuropsychological Status (RBANS) - Attention Digit Span - day 8, admin 1 | During the evening cognitive testing on Overnight Visit 1 (day 8)
  To measure auditory registration and attention. The examiner reads aloud a set of numbers and asks the participant to repeat them back to them. The examinee repeats them back verbally. Participant is scored based on correctly repeating back the string of numbers (2 points for getting it right on the first trial using the Repeatable Battery for the Assessment of Neuropsychological Status Attention Digit Span scale (0-16, higher number indicates better outcome)
Repeatable Battery for Neuropsychological Status (RBANS) - Attention Digit Span - day 15, admin 1 | During the evening cognitive testing on Overnight Visit 2 (day 15)
  To measure auditory registration and attention. The examiner reads aloud a set of numbers and asks the participant to repeat them back to them. The examinee repeats them back verbally. Participant is scored based on correctly repeating back the string of numbers (2 points for getting it right on the first trial using the Repeatable Battery for the Assessment of Neuropsychological Status Attention Digit Span scale (0-16, higher number indicates better outcome).
Repeatable Battery for Neuropsychological Status (RBANS) - Attention Digit Span - day 9, admin 2 | During the morning cognitive testing on Overnight Visit 1 (day 9)
  To measure auditory registration and attention. The examiner reads aloud a set of numbers and asks the participant to repeat them back to them. The examinee repeats them back verbally. Participant is scored based on correctly repeating back the string of numbers (2 points for getting it right on the first trial using the Repeatable Battery for the Assessment of Neuropsychological Status Attention Digit Span scale (0-16, higher number indicates better outcome).
Repeatable Battery for Neuropsychological Status (RBANS) - Attention Digit Span - day 16, admin 2 | During the morning cognitive testing on Overnight Visit 2 (day 16)
  To measure auditory registration and attention. The examiner reads aloud a set of numbers and asks the participant to repeat them back to them. The examinee repeats them back verbally. Participant is scored based on correctly repeating back the string of numbers (2 points for getting it right on the first trial using the Repeatable Battery for the Assessment of Neuropsychological Status Attention Digit Span scale (0-16, higher number indicates better outcome).
Repeatable Battery for Neuropsychological Status (RBANS) - Delayed Memory Story Recall - day 8, admin 1 | During the evening cognitive testing on Overnight Visit 1 (day 8)
  To measure delayed recall and recognition for verbal information.The examiner reads a short story aloud to the participant, then later, the participant is asked to recall the story in as much detail as possible. Participant is scored based on the number of units of information correctly recalled using the Repeatable Battery for the Assessment of Neuropsychological Status Delayed Story Memory scale (0-12, higher number indicates better outcome).
Repeatable Battery for Neuropsychological Status (RBANS) - Story Memory Recall - day 8 | During the evening cognitive testing on Overnight Visit 1 (day 8)
  To measure delayed recall and recognition for verbal information. The examiner reads a short story aloud to the participant and then the participant is asked to recall the story in as much detail as possible. This is repeated twice. The Participant is scored based on the number of units of information correctly recalled using the Repeatable Battery for the Assessment of Neuropsychological Status Story Memory scale (0-24, higher number indicates better outcome).
Repeatable Battery for Neuropsychological Status (RBANS) - Delayed Memory Story Recall - day 15, admin 1 | During the evening cognitive testing on Overnight Visit 2 (day 15)
  To measure delayed recall and recognition for verbal information.The examiner reads a short story aloud to the participant, then later, the participant is asked to recall the story in as much detail as possible. Participant is scored based on the number of units of information correctly recalled using the Repeatable Battery for the Assessment of Neuropsychological Status Delayed Story Memory scale (0-12, higher number indicates better outcome).
Repeatable Battery for Neuropsychological Status (RBANS) - Story Memory Recall - day 15 | During the evening cognitive testing on Overnight Visit 2 (day 15)
  To measure delayed recall and recognition for verbal information. The examiner reads a short story aloud to the participant and then the participant is asked to recall the story in as much detail as possible. This is repeated twice. The Participant is scored based on the number of units of information correctly recalled using the Repeatable Battery for the Assessment of Neuropsychological Status Story Memory scale (0-24, higher number indicates better outcome).
Repeatable Battery for Neuropsychological Status (RBANS) - Delayed Memory Story Recall - day 9, admin 2 | During the morning cognitive testing on Overnight Visit 1 (day 9)
  To measure delayed recall and recognition for verbal information.The examiner reads a short story aloud to the participant, then later, the participant is asked to recall the story in as much detail as possible. Participant is scored based on the number of units of information correctly recalled using the Repeatable Battery for the Assessment of Neuropsychological Status Delayed Story Memory scale (0-12, higher number indicates better outcome).
Repeatable Battery for Neuropsychological Status (RBANS) - Delayed Memory Story Recall - day 16, admin 2 | During the morning cognitive testing on Overnight Visit 2 (day 16)
  To measure delayed recall and recognition for verbal information.The examiner reads a short story aloud to the participant, then later, the participant is asked to recall the story in as much detail as possible. Participant is scored based on the number of units of information correctly recalled using the Repeatable Battery for the Assessment of Neuropsychological Status Delayed Story Memory scale (0-12, higher number indicates better outcome).
Repeatable Battery for Neuropsychological Status (RBANS) - Symbol-Digit Test - day 8, admin 1 | During the evening cognitive testing on Overnight Visit 1 (day 8)
  To assess tracking and motor speed, divided attention, and visual scanning. Participants will be given a simple substitution task to pair specific numbers with provided geometric figures. Participant is scored based on the number of correct answers using the Repeatable Battery for the Assessment of Neuropsychological Status Symbol-Digit scale (0-89, higher number indicates better outcome).
Repeatable Battery for Neuropsychological Status (RBANS) - Symbol-Digit Test - day 15, admin 1 | During the evening cognitive testing on Overnight Visit 2 (day 15)
  To assess tracking and motor speed, divided attention, and visual scanning. Participants will be given a simple substitution task to pair specific numbers with provided geometric figures. Participant is scored based on the number of correct answers using the Repeatable Battery for the Assessment of Neuropsychological Status Symbol-Digit scale (0-89, higher number indicates better outcome).
Repeatable Battery for Neuropsychological Status (RBANS) - Symbol-Digit Test - day 9, admin 2 | During the morning cognitive testing on Overnight Visit 1 (day 9)
  To assess tracking and motor speed, divided attention, and visual scanning. Participants will be given a simple substitution task to pair specific numbers with provided geometric figures. Participant is scored based on the number of correct answers using the Repeatable Battery for the Assessment of Neuropsychological Status Symbol-Digit scale (0-89, higher number indicates better outcome).
Repeatable Battery for Neuropsychological Status (RBANS) - Symbol-Digit Test - day 16, admin 2 | During the morning cognitive testing on Overnight Visit 2 (day 16)
  To assess tracking and motor speed, divided attention, and visual scanning. Participants will be given a simple substitution task to pair specific numbers with provided geometric figures. Participant is scored based on the number of correct answers using the Repeatable Battery for the Assessment of Neuropsychological Status Symbol-Digit scale (0-89, higher number indicates better outcome).
Visual Attention Task (VAT) - day 8, admin 1 | Once during pre-TMS MRI scan on evening of Overnight Visit 1 (day 8)
  To assess default mode network connectivity during a visual attention task. While inside the 3T scanner, participants will identify global and local letters from visually presented stimuli. This task will be administered pre-TMS and trials will be randomized to prevent task habituation. Participant is scored based on the number of correct responses they provide (0-192, higher number indicates better outcome).
Visual Attention Task (VAT) - day 8, admin 2 | Once during post-TMS MRI scan on evening of Overnight Visit 1 (day 8)
  To assess default mode network connectivity during a visual attention task. While inside the 3T scanner, participants will identify global and local letters from visually presented stimuli. This task will be administered post-TMS and trials will be randomized to prevent task habituation. Participant is scored based on the number of correct responses they provide (0-192, higher number indicates better outcome).
Visual Attention Task (VAT) - day 15, admin 1 | Once during pre-TMS MRI scan on evening of Overnight Visit 2 (day 15)
  To assess default mode network connectivity during a visual attention task. While inside the 3T scanner, participants will identify global and local letters from visually presented stimuli. This task will be administered pre-TMS and trials will be randomized to prevent task habituation. Participant is scored based on the number of correct responses they provide (0-192, higher number indicates better outcome).
Visual Attention Task (VAT) - day 15, admin 2 | Once during post-TMS MRI scan on evening of Overnight Visit 2 (day 15)
  To assess default mode network connectivity during a visual attention task. While inside the 3T scanner, participants will identify global and local letters from visually presented stimuli. This task will be administered post-TMS and trials will be randomized to prevent task habituation. Participant is scored based on the number of correct responses they provide (0-192, higher number indicates better outcome).
Multi-Source Interference Task (MSIT) - day 8, admin 1 | Once during pre-TMS scan on evening of Overnight Visit 1 (day 8)
  To assess default mode network connectivity during a visual interference task. Use index, middle, or ring finger to press button that indicates the spatial location of the "number 1" on the screen. In the "interference" condition, participants will see three numbers, two of which are the same, and they will use the same buttons to choose the number that is different. This is administered pre-TMS.
Multi-Source Interference Task (MSIT) - day 8, admin 2 | Once during post-TMS scan on evening of Overnight Visit 1 (day 8)
  To assess default mode network connectivity during a visual interference task. Use index, middle, or ring finger to press button that indicates the spatial location of the "number 1" on the screen. In the "interference" condition, participants will see three numbers, two of which are the same, and they will use the same buttons to choose the number that is different. This is administered post-TMS.
Multi-Source Interference Task (MSIT) - day 15, admin 1 | Once during pre-TMS scan on evening of Overnight Visit 2 (day 15)
  To assess default mode network connectivity during a visual interference task. Use index, middle, or ring finger to press button that indicates the spatial location of the "number 1" on the screen. In the "interference" condition, participants will see three numbers, two of which are the same, and they will use the same buttons to choose the number that is different. This is administered pre-TMS.
Multi-Source Interference Task (MSIT) - day 15, admin 2 | Once during post-TMS scan on evening of Overnight Visit 2 (day 15)
  To assess default mode network connectivity during a visual interference task. Use index, middle, or ring finger to press button that indicates the spatial location of the "number 1" on the screen. In the "interference" condition, participants will see three numbers, two of which are the same, and they will use the same buttons to choose the number that is different. This is administered post-TMS.

CONTACTS AND LOCATIONS:
Overall Officials: William D Killgore, PhD, Principal Investigator — University of Arizona
Locations (1):
- University of Arizona Psychiatry Department, Tucson, Arizona, United States

REFERENCES:
- [Derived] Huskey A, Fisher JM, Hildebrand L, Negelspach D, Henderson-Arredondo K, Jankowski S, Patel SI, Chou YH, Dailey NS, Killgore WDS. Polysomnographically mediated cognitive improvements in individuals with insomnia symptoms following continuous theta-burst stimulation of the default mode network. Front Sleep. 2024 Oct 2;3:1424083. doi: 10.3389/frsle.2024.1424083. eCollection 2024. PMID 41424521
- [Derived] Hildebrand L, Huskey A, Dailey N, Jankowski S, Henderson-Arredondo K, Trapani C, Patel SI, Chen AY, Chou YH, Killgore WDS. Transcranial Magnetic Stimulation of the Default Mode Network to Improve Sleep in Individuals With Insomnia Symptoms: Protocol for a Double-Blind Randomized Controlled Trial. JMIR Res Protoc. 2024 Jan 26;13:e51212. doi: 10.2196/51212. PMID 38277210